CLINICAL TRIAL: NCT05244954
Title: Clinical Trial to Evaluate Intermittent Screening and Treatment and Intermittent Preventive Treatment of Malaria in Asymptomatic Schoolchildren to Decrease P. Falciparum Infection and Transmission
Brief Title: Comparing Chemoprevention Approaches for School-based Malaria Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Lauren Cohee, Visiting Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00098250
Record Dates: First submitted 2022-01-11; First posted 2022-02-17 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Malaria,Falciparum; Anemia in Children
Keywords: malaria; school; chemoprevention; preventive treatment; screening and treatment; education; cognitive function; adolescent; hemoglobin
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Chloroquine

STUDY DESIGN:
Intervention Model Description: Students will be randomized to intermittent screening-and-treatment (IST - Arm 1), intermittent preventive treatment (IPT - Arm 2), or control with no preventive treatment (Arm 3). Females less that 10 years of age (pre-menarche) and all males will be treated with DP if they are in Arm 2 or test positive in Arm 1. Females 10 years and older will be treated with chloroquine if they are in Arm 2 or test positive in Arm 1.
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians processing samples will be blinded to participant's study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent Screening and Treatment (IST) (Experimental): Students will be screened for infection using a higher sensitivity malaria rapid diagnostic test and treated if positive. Treatment will be with DP (females less than 10 years old and all males) or chloroquine (females 10 years old or older).
  Interventions: Drug: Dihydroartemisinin-Piperaquine; Drug: Chloroquine
- Intermittent Preventive Treatment (IPT) (Experimental): All students are treated at each intervention. Treatment will be with DP (females less than 10 years old and all males) or chloroquine (females 10 years old or older).
  Interventions: Drug: Dihydroartemisinin-Piperaquine; Drug: Chloroquine
- Control (No Intervention): Students will not receive preventive treatment.

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine — Treatment of females less than 10 years old and all males in Arm 2 and those who test positive in Arm 1.
  Other Names: DP; DuoCotecxin; Artekin; Eurartesim; Ridmal
  Arms: Intermittent Preventive Treatment (IPT); Intermittent Screening and Treatment (IST)
Drug: Chloroquine — Treatment of females 10 years old and older in Arm 2 and those who test positive in Arm 1.
  Other Names: Aralen
  Arms: Intermittent Preventive Treatment (IPT); Intermittent Screening and Treatment (IST)

SUMMARY:
This is an individually randomized, controlled, single blind three arm clinical trial of malaria chemoprevention strategies Arm 1: Intermittent screening and treatment (IST) - students will receive treatment if they have a positive high sensitivity rapid diagnostic test (RDT). Arm 2: Intermittent preventive treatment (IPT) - all students will receive treatment. Arm 3: Control - students will receive standard of care (no preventive treatment). Outcomes include P. falciparum infection and parasite density, gametocyte carriage and gametocyte density, anemia, cognitive function and educational testing, as well as infection prevalence in student's households to assess the impact on transmission.

DETAILED DESCRIPTION:
Students will be enrolled in a single primary school in Machinga District, Malawi. The intervention will be conducted every 6-weeks during the two school terms which coincide with peak malaria transmission. Students in the IPT are and those that test positive in the IST arm will be treatment with dihydroartemisinin-piperaquine (DP) (females less than 10 years old and all males) or chloroquine (females 10 years old or older).

ELIGIBILITY:
Inclusion Criteria:

Students (enrolled in the primary intervention)

* Currently enrolled in the study school
* Plan to attend the study school for the remainder of the school year
* Parent/guardian available to provide written informed consent Household members (enrolled in the Household Prevalence survey)
* Slept in the household for most nights in the last month
* Age 6 months or older
* For minors, parent/guardian available to provide written informed consent

Exclusion Criteria:

Students (enrolled in the primary intervention)

* Current evidence of severe malaria or danger signs
* Known adverse reaction to the study drugs
* History of cardiac problems or fainting
* Taking medications known to prolong QT
* Family history of prolonged QT
* Girls 10 years old and older with epilepsy or psoriasis Household members (enrolled in the Household Prevalence survey)
* Household with more than one school-age child enrolled in the study
* Current evidence of severe malaria or danger signs

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
P. falciparum infection | 6-8 weeks after the last intervention
  detected by polymerase chain reaction (PCR, binary)
P. falciparum gametocyte carriage | 6-8 weeks after the last intervention
  detected by q-rtPCR (binary)

SECONDARY OUTCOMES:
Number of participant with anemia | 6-8 weeks after the last intervention
  World Health Organization age-sex definitions (binary)
Mean hemoglobin concentration | 6-8 weeks after the last intervention
  g/dL (continuous)
Total parasite density | 6-8 weeks after the last intervention
  log transformed (continuous)
Gametocyte density | 6-8 weeks after the last intervention
  log transformed (continuous)
Rate of clinical malaria | from the first intervention to 6-8 weeks after the last intervention
  cumulative incidence
P. falciparum prevalence among household members | 6-8 weeks after the last intervention
  detected by PCR

OTHER OUTCOMES:
Cognitive function test scores | 6-8 weeks after the last intervention
  standardized scores
Reading test scores | 6-8 weeks after the last intervention
  standardized scores
Math test scores | 6-8 weeks after the last intervention
  standardized scores
School attendance | from the first intervention to 6-8 weeks after the last intervention
  number of days missed based on registers and spot checks
Mean infectiousness | from the first intervention to 6-8 weeks after the last intervention
  regression modeled infectiousness based on gametocyte density, gametocyte sex ratio, symptom status, and other predictors of infectiousness
Performance characteristics of conventional RDT | through study completion, on average 6 months
  compared to PCR to detect: P. falciparum infection, P. falciparum parasite density, anemia, hemoglobin, gametocytemia, gametocyte density, and potential infectiousness score
Performance characteristics of high-sensitivity RDT | through study completion, on average 6 months
  compared to PCR to detect: P. falciparum infection, P. falciparum parasite density, anemia, hemoglobin, gametocytemia, gametocyte density, and potential infectiousness score

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Cohee, MD MS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Kamuzu University of Health Sciences, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After results publication
Access Criteria: Public access with registration to allow tracking

REFERENCES:
- [Background] Cohee LM, Valim C, Coalson JE, Nyambalo A, Chilombe M, Ngwira A, Bauleni A, Seydel KB, Wilson ML, Taylor TE, Mathanga DP, Laufer MK. School-based screening and treatment may reduce P. falciparum transmission. Sci Rep. 2021 Mar 25;11(1):6905. doi: 10.1038/s41598-021-86450-5. PMID 33767384
- [Background] Cohee LM, Opondo C, Clarke SE, Halliday KE, Cano J, Shipper AG, Barger-Kamate B, Djimde A, Diarra S, Dokras A, Kamya MR, Lutumba P, Ly AB, Nankabirwa JI, Njagi JK, Maiga H, Maiteki-Sebuguzi C, Matangila J, Okello G, Rohner F, Roschnik N, Rouhani S, Sissoko MS, Staedke SG, Thera MA, Turner EL, Van Geertruyden JP, Zimmerman MB, Jukes MCH, Brooker SJ, Allen E, Laufer MK, Chico RM. Preventive malaria treatment among school-aged children in sub-Saharan Africa: a systematic review and meta-analyses. Lancet Glob Health. 2020 Dec;8(12):e1499-e1511. doi: 10.1016/S2214-109X(20)30325-9. Epub 2020 Oct 22. PMID 33222799
- [Background] Halliday KE, Okello G, Turner EL, Njagi K, Mcharo C, Kengo J, Allen E, Dubeck MM, Jukes MC, Brooker SJ. Impact of intermittent screening and treatment for malaria among school children in Kenya: a cluster randomised trial. PLoS Med. 2014 Jan 28;11(1):e1001594. doi: 10.1371/journal.pmed.1001594. eCollection 2014 Jan. PMID 24492859